CLINICAL TRIAL: NCT03771573
Title: Physical Therapy in Rehabilitation Program on Cardiovascular Diseases
Brief Title: Rehabilitation With Exercises in Cardiovascular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Collaborators: Universidade do Estado do Pará (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, Principal invastigator, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2.728.401
Record Dates: First submitted 2018-12-03; First posted 2018-12-11 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Diseases
Keywords: REHABILITATION; PHYSICAL THERAPY; CARDIOVASCULAR DISEASE
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: BLINDED AND RANDOMIZED CLINICAL TRIAL
Who Masked: Investigator
Masking Description: THE BLIND INVESTIGATOR, WHO WILL NOT KNOW THE GROUPS AND THE STUDY, WILL RECEIVE THE DATED NAMES WITH CODES TO CARRY OUT DATA ANALYSIS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home based intervention (Experimental): will be submitted to a total of 24 sessions of an unsupervised Cardiovascular Physical Therapy protocol, composed of the following steps: warm up, proper training (aerobic training + muscle training for upper and lower limbs with theraband in 5 series with 10 repetitions) often three times a week for eight weeks.
  Interventions: Other: Physical exercise
- Control group (Placebo Comparator): Will not be submitted to the Cardiovascular Physiotherapy Rehabilitation protocol for unsupervised domiciliary, only monitorization of cardiovascular variables.
  Interventions: Other: monitoring
- Professional seupervision based (Active Comparator): eight weeks of supervised activities by professional. Each day and for 20 days (20 sessions), volunteers will undergo exercises on cycle ergometer during 30 minutes for upper and lower limbs
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — Participants will perform physical exercises with constant, or intermittent professional supervision or will interrupt the exercise after ambulatorial physical therapy
  Arms: Home based intervention; Professional seupervision based
Other: monitoring — the patients will be under monitoring to investigate the evolution of the disease
  Arms: Control group

SUMMARY:
INTRODUCTION: Cardiovascular diseases are the main causes of death in Brazil and in the world, associated with a large number of people with physical disabilities and disability, significantly burdening public health expenditures. Some patients end up having the need to do cardiac surgeries. , and consequently suffer complications associated with the surgical process due to prolonged rest in the bed, and complications are directly related to the morbidity and mortality rate in these patients. Thus, cardiac rehabilitation has great scientific evidences that directly impacts functional capacity, quality of life and thus reducing the morbimortality rate of these patients. However, it is worth noting that there is no outpatient cardiovascular rehabilitation service linked to the single health system (SUS) in the Amazon Region, that is, involving phase III of cardiac rehabilitation with defined and structured protocols for the group of patients already mentioned. OBJECTIVE: To analyze the clinical evolution of patients in the postoperative period of coronary artery bypass grafting and / or valve replacement (phase III), in outpatient treatment. METHODOLOGY: It is a a longitudinal study, with quantitative variables to be performed in a single center within a year (12 months). Which will evaluate the effects of phase III cardiac rehabilitation of patients undergoing cardiac surgery through an evaluation, which will evaluate heart rate variability, functional capacity by six-minute walk test, pulmonary volumes and capacities by spirometry, percutaneous strength and ventilatory muscle, MRC scale and manovacuometry, respectively, and the application of a quality of life assessment questionnaire. Subsequently, the protocol of 20 sessions will be applied and at the end the same variables will be re-evaluated. EXPECTED RESULTS: It is expected from the application of this research that the protocol suggested for the phase III cardiac rehabilitation of patients submitted to cardiac surgery will bring benefits to patients, such as improvement in heart rate variability, improvement in functional capacity, improvement in quality of life, and reduction in morbidity and mortality rates.

DETAILED DESCRIPTION:
Characterized by the insufficiency of blood supply to the heart through the coronary arteries, coronary artery disease (CAD) stands out as a global health problem, since it represents the main cause of morbidity and mortality and is among the pathologies with the greatest clinical and significantly increasing public health expenditures. In Brazil, it is estimated that CAD corresponds to 80% of deaths due to cardiovascular diseases (CVD), mainly in large centers and in the population with age over 40 years. CAD is associated with risk factors such as systemic arterial hypertension, smoking, dyslipidemia, obesity, diabetes mellitus, sedentary lifestyle, and in addition to the family history of coronary insufficiency, that favors its onset.

The process of treatment of CAD is variable according to the level of involvement, and can be performed through drugs, physical activities, nutritional control and surgical procedure. Cardiac surgery is an alternative to promote improvement of cardiovascular function in addition to reduction of morbimortality rates due to circulatory diseases, only performed when clinical treatment is not able to provide cure and / or improvement of patient's quality of life. Myocardial revascularization (CABG) surgery is one of the most accomplished cardiac surgeries in Brazil, and it is currently recognized as a well-established procedure for the treatment of CAD, since it is capable of prolonging and improving the quality of life of these patients.

CABG aims at the resolution of myocardial ischemia, seeking the relief of symptoms and consequently improvement of patient survival, biopsychosocial well-being, as well as the earlier return to their daily activities, however, because it is an invasive procedure and complexity, can imply several systemic repercussions such as cardiac, renal, infectious, motor and pulmonary alterations. The postoperative complications of CABG depend on factors related to the clinical situation at the time of surgery, such as age, life habits, comorbidities, and also factors associated with the surgical process, such as duration of surgery, use of extracorporeal circulation, schedules and the long-term invasive mechanical ventilation and hospitalization.

Respiratory complications after CABG contribute to the reduction of the patients' quality of life and increased morbimortality rates. Decreased respiratory muscle strength may be a result of respiratory muscle injury during surgery and / or secondary to diaphragmatic dysfunction due to phrenic nerve injury. Respiratory muscle weakness may compromise the ventilation structure and function of these patients, exacerbating dyspnea, effort intolerance, decreased ability to perform physical exercise, and consequently reduced functional capacity (FC) of the individuals. The FC has a direct impact on the performance of activities of daily living (ADLs), and in this context, the practice of physical exercise after cardiac surgery is essential in the functional recovery of patients.

Cardiovascular rehabilitation (CVR) has a "1" level of recommendation and "A" grade of scientific evidence, and physiotherapy has been the main component in this process, being strongly associated with increased exercise capacity, improved dyspnea, quality of life, as well as a decrease in mortality and morbidity rates, leading to an increase in the life expectancy of these patients in the postoperative period .

Despite the well-known benefits of CVR, the number of patients participating in this program is considered small, only 34% of the candidates are targeted and in the end, only 20% of these candidates participate. In addition, as regards Phase IV rehabilitation, health management of patients is still limited as improvements in lifestyle behavior are often not maintained in the long run and levels of physical activity generally decline after a program of successful outpatient rehabilitation, resulting in the loss of adaptations acquired as a result of physical training.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery;
* Both sexes and age group between 40 and 70 years;
* Who were discharged from ambulatory;
* That they agree to participate in the survey

Exclusion Criteria:

* Patients with Osteomioarticular diseases in upper and lower limbs and neurological diseases that may interfere with the performance of the exercises proposed in the protocol.
* Female patients in the climacteric.
* Patients with cardiovascular diseases such as uncontrolled arterial hypertension, arrhythmias that use cardiac pacemakers, infectious diseases that affect the cardiovascular system such as Chagas disease, Heart Failure and / or patients with diabetes mellitus.
* With simultaneous lung diseases, such as asthma, COPD, collagen diseases (eg, scleroderma) and sarcoidosis.
* Occupational diseases, such as pneumoconiosis, hypersensitivity pneumonia.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | during 3 months
  For the collection, the patients will be placed in the supine position and kept at rest for 10 minutes to stabilize the vital signs, after which HR and RR intervals (iR-R) will be recorded, with a duration of 10 minutes. Patient oriented not to perform movements and not to talk during the collection period.
  The recording of the VFC will be performed by means of a POLAR® brand, RS800CX (Polar Electro TM, Kempele, Finland), where the HR signal will be picked up by a strap with the signal receiver placed in the patient's chest at the time of the xiphoid process of the sternum.
  The data recorded by the frequency meter will be transferred to the Polar ProTrainer® Software via an infrared signal emitting interface, where it will be stored and subsequently exported in .txt format.
  The data obtained will be compared before and after the completion of the cardiovascular rehabilitation protocol in the control and intervention groups, among the same.
Respiratoey muscle strenght | during 3 months
  Respiratory muscle strength is evaluated with a digital manovacuometer. The patient in the seated position and using a nasal clip performs up to eight maximal inspiration and expiration maneuvers. Measurement of MIP occurs as follows: a nasal clip is used to prevent air from escaping through the nostrils and patients are instructed to place the connection mouthpiece to the manometer, then it is required to empty the lungs. The highest recorded value is the one used for the analysis. In order to measure PEmáx, the patient is asked to fill the air lungs as far as possible to the CPT, making a forced inspiration, and then, with the nasal clip and the manovacuometer connection nozzle correctly positioned, to perform an expiration up to the VR level, held for one second. This maneuver is also performed three times and its values were recorded by the equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo S Rocha, Phd, Principal Investigator — Universidade do Estado do Pará
Locations (1):
- Universidade da Amazônia, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Anderson L, Oldridge N, Thompson DR, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-Based Cardiac Rehabilitation for Coronary Heart Disease: Cochrane Systematic Review and Meta-Analysis. J Am Coll Cardiol. 2016 Jan 5;67(1):1-12. doi: 10.1016/j.jacc.2015.10.044. PMID 26764059
- [Result] Borges JP, Mediano MF, Farinatti P, Coelho MP, Nascimento PM, Lopes GO, Kopiler DA, Tibirica E. The Effects of Unsupervised Home-based Exercise Upon Functional Capacity After 6 Months of Discharge From Cardiac Rehabilitation: A Retrospective Observational Study. J Phys Act Health. 2016 Nov;13(11):1230-1235. doi: 10.1123/jpah.2016-0058. Epub 2016 Aug 24. PMID 27333938
- [Result] Lavie CJ, Arena R, Swift DL, Johannsen NM, Sui X, Lee DC, Earnest CP, Church TS, O'Keefe JH, Milani RV, Blair SN. Exercise and the cardiovascular system: clinical science and cardiovascular outcomes. Circ Res. 2015 Jul 3;117(2):207-19. doi: 10.1161/CIRCRESAHA.117.305205. PMID 26139859
- [Result] Caruso FC, Simoes RP, Reis MS, Guizilini S, Alves VL, Papa V, Arena R, Borghi-Silva A. High-Intensity Inspiratory Protocol Increases Heart Rate Variability in Myocardial Revascularization Patients. Braz J Cardiovasc Surg. 2016 Feb;31(1):38-44. doi: 10.5935/1678-9741.20160007. PMID 27074273
- [Result] Hamm LF, Wenger NK, Arena R, Forman DE, Lavie CJ, Miller TD, Thomas RJ. Cardiac rehabilitation and cardiovascular disability: role in assessment and improving functional capacity: a position statement from the American Association of Cardiovascular and Pulmonary Rehabilitation. J Cardiopulm Rehabil Prev. 2013 Jan-Feb;33(1):1-11. doi: 10.1097/HCR.0b013e31827aad9e. PMID 23254246